CLINICAL TRIAL: NCT00467948
Title: Double Blind Randomised Study of 2 Days and 5 Days Cefazolin Prophylactic Method in Laryngeal Oncologic Surgery
Brief Title: Comparison of 2 Cefazolin Prophylactic Protocol in Laryngectomy Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BS_200306
Record Dates: First submitted 2007-04-29; First posted 2007-05-01 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2003-06

CONDITIONS: Laryngeal Cancer
Keywords: clean contaminated, laryngectomy, wound infection
MeSH Terms: conditions — Laryngeal Neoplasms; Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cefazolin

SUMMARY:
Patients who need major head & neck surgery are at risk of post operative wound infection. In spite of role of antibiotics in prophylaxis of clean contaminated head and neck surgery has been well documented, controversy exists in the optimal antibiotic regimen

DETAILED DESCRIPTION:
Patients undergoing laryngeal oncologic surgery are at relatively high risk of developing complication.

Efficacy of cefazolin as a prophylactic antibiotic in head and neck surgery was reviewed in many researches [6] but considering the costs and morbidities of prolonged antibiotic regimen we have presented a prospective and randomized study in 90 patients comparing the efficacy of 2 day over 5 day protocols.

ELIGIBILITY:
Inclusion Criteria:e.

* Patients eligible to be included in this trial were those who histologically confirmed squamous cell carcinoma of larynx and hypopharynx and they were candidate of total or partial laryngectomy with or without neck dissection and with negative history of neck or laryngeal radiation were included in this study.

Exclusion Criteria:

* Patients having recurrences or another primary tumor, and those who underwent reconstruction with a flap were excluded from the study, because they had been submitted to prolonged antibiotic administration. Also cases with Diabet mellitus and Immune suppression or tumor types other than squamous cell carcinoma were excluded from the study.
* In addition, the following exclusion criteria were taken into account: pregnancy, hypersensitivity to penicillins or cephalosporins, patients who received a systemic antibiotic drug within one week prior to the planned procedure, those who had clinical or laboratory evidence of a preexisting infection or had serious systemic renal disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-06; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
wound infection | prospective

SECONDARY OUTCOMES:
drug complication | 3 week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: taghi khorsandi, professor, Study Chair — tehran university of medical science
Locations (1):
- Imam khomaini hospital, Tehran, Tehran Province, Iran